CLINICAL TRIAL: NCT01752751
Title: Predicting Tolerance to Radiation Therapy in Older Adults With Cancer: A Prospective Blinded Study of the Comprehensive Geriatric Assessment
Brief Title: Predicting Tolerance to Radiation Therapy in Older Adults With Cancer
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Alpha Omega Alpha Honor Medical Society (Unknown)
Responsible Party: Sponsor
Other Study IDs: LCCC 1224; 1224 (Other Grant/Funding Number: Lineberger Cancer Center); 121731 (Other: UNC IRB)
Record Dates: First submitted 2012-12-14; First posted 2012-12-19 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Pre-treatment Loss of Independent Activities of Daily Living
Keywords: Neck cancer; Head cancer; Lung cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cancer Patients Age 65 or above: Cancer patients age 65 years or above with a diagnosis of head and neck cancer or lung cancer with radiotherapy or chemoradiotherapy planned as part of curative standard treatment.

SUMMARY:
A comprehensive geriatric assessment tool developed by Hurria and colleagues has been used in non-radiation oncology clinical settings to predict how older adults tolerate cancer treatments. The investigators think this same tool (referred to as the CGA) can be used in a radiation oncology clinic to predict for poor treatment tolerance.

DETAILED DESCRIPTION:
A comprehensive geriatric assessment tool developed by Hurria and colleagues has been used in non-radiation oncology clinical settings to predict for toxicity in older patients during cancer treatments.1 The investigators hypothesize that the same tool (referred to throughout this document as the CGA) can be used in a radiation oncology clinic to predict for poor treatment tolerance. The primary objective of this study is to assess the association between pre-treatment functional status (as measured by the Independent Activities of Daily Living (I-ADL) components of the CGA) and poor tolerance to radiation therapy (as defined in section 2.3.1). Secondary objectives include exploration of associations between pre-treatment I-ADL status on the CGA and the occurrence of any acute grade 3-5 toxicity from radiation therapy, or any decrease in Quality of Life (QoL) measures throughout radiation therapy as assessed by the EORTC QLQ-C30 questionnaire. The investigators also want to compare the rate of physician reported acute toxicities to patient reported acute toxicities in an older cancer patient population, assess any association between elevated p16Ink4α expression in peripheral T lymphocytes and poor tolerance to or acute grade 3-5 toxicity from radiation therapy, and explore any association between other baseline components of the CGA and poor tolerance to or acute grade 3-5 toxicity from radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* ≥Age 65 years (no upper age limit)
* Diagnosis of either head and neck cancer, or lung cancer with either radiotherapy or chemoradiotherapy planned as part of standard treatment.
* Consented for receipt of External Beam Radiation Therapy (EBRT) at UNC Chapel Hill
* Able to read English (required for CGA)
* Curative treatment intent as defined by their radiation oncologist Signed, IRB-approved written informed consent
* Patients enrolled in other CGA studies will not be excluded (see LCCC 0916, 1208)

Exclusion Criteria:

* ≥Age 65 years (no upper age limit)
* Diagnosis of either head and neck cancer, or lung cancer with either radiotherapy or chemoradiotherapy planned as part of standard treatment.
* Consented for receipt of EBRT at UNC Chapel Hill
* Able to read English (required for CGA)
* Curative treatment intent as defined by their radiation oncologist Signed, IRB-approved written informed consent
* Patients enrolled in other CGA studies will not be excluded (see LCCC 0916, 1208)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients age ≥ 65 years of age, with one of the inclusion diagnoses, and an appointment for CT simulation for planning of radiation therapy at UNCH department of radiation oncology will be assessed for inclusion for this study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Association between pre-treatment loss of at least one independent activity of daily living (I-ADL) and poor tolerance to radiation therapy | 4-8 weeks post-radiation therapy
  To assess the association between pre-treatment loss of at least one independent activity of daily living (I-ADL) on the CGA and poor tolerance to radiation therapy

SECONDARY OUTCOMES:
Association between pre-treatment loss of at least one independent activity of daily living (I-ADL) and the occurrence of any patient-reported toxicity from radiation therapy | 4-8 weeks post-radiation therapy
  To assess the association between pre-treatment loss of at least one I-ADL on the CGA and the occurrence of any patient-reported acute grade 3-5 toxicity from radiation therapy
Association between pre-treatment loss of at least one independent activity of daily living and changes in Quality of Life measures | 4-8 weeks post radiation therapy
  To assess the association between pre-treatment loss of at least one I-ADL on the CGA and changes in QoL measures, as evaluated by the EORTC-QLQ-C30 throughout radiation therapy
Comparison of physician and patient-reported acute grade 3-5 toxicities | 4-8 weeks post-radiation therapy
  To compare physician-reported acute grade 3-5 toxicities to patient-reported grade 3-5 acute toxicities in this older adult population.
Association between elevated p16Ink4α gene expression and poor tolerance to and/or physician/patient-reported toxicity from radiation therapy | 4-8 weeks post-radiation therapy
  To assess the association between elevated p16Ink4α expression in peripheral T lymphocytes and poor tolerance to and/or patient reported and physician reported acute grade 3-5 toxicity from radiation therapy
Association between baseline components of the Comprehensive Geriatric Assessment and poor tolerance to or occurrence of patient-reported toxicity from radiation treatment | 4-8 weeks post-radiation therapy
  To explore the association between baseline components of the CGA (other than I-ADL) and poor tolerance to or occurrence of any patient-reported acute grade 3-5 toxicity from radiation treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Bhishamjit Chera, MD, Principal Investigator — Radiation Oncology UNC Cancer Hospital; Noam VanderWalde, MD, Study Director — Radiation Oncology UNC Cancer Hospital
Locations (1):
- Radiation Oncology Clinic - UNC Cancer Hospital, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] VanderWalde NA, Deal AM, Comitz E, Stravers L, Muss H, Reeve BB, Basch E, Tepper J, Chera B. Geriatric Assessment as a Predictor of Tolerance, Quality of Life, and Outcomes in Older Patients With Head and Neck Cancers and Lung Cancers Receiving Radiation Therapy. Int J Radiat Oncol Biol Phys. 2017 Jul 15;98(4):850-857. doi: 10.1016/j.ijrobp.2016.11.048. Epub 2016 Dec 2. PMID 28258889